CLINICAL TRIAL: NCT03473340
Title: A Phase Two Randomized, Double-blinded, Placebo-controlled Study Combining Physiological, Radiographic, and Biological Biomarkers to Study the Anti-fibrotic Effect of Pirfenidone in CLAD Post Lung-transplantation
Brief Title: Studying the Treatment Effect of Pirfenidone in Chronic Lung Allograft Dysfunction (STOP-CLAD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow and delayed recruitment due in part to COVID, led to a decision to end funding and terminate the trial.
Sponsor: University of Michigan (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Vibha Lama, Henry Sewall Research Professor of Pulmonary and Critical Care Medicine and Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00131610
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Results first posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-07

CONDITIONS: Disorder Related to Lung Transplantation; Chronic Lung Allograft Dysfunction
Keywords: CLAD; Chronic Rejection; Lung Transplant
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pirfenidone Capsule (Experimental): Method of Administration: Oral (capsule)
  Dosing:
  * Days 1 through 7, 267 mg three times daily;
  * Days 8 through 14, 534 mg three times daily;
  * Days 15 through end of treatment (24 weeks), 801 mg three times daily
  Interventions: Drug: Pirfenidone Capsule
- Placebo Capsule (Placebo Comparator): Method of Administration: Oral (capsule)
  Dosing:
  * Days 1 through 7, 267 mg three times daily;
  * Days 8 through 14, 534 mg three times daily;
  * Days 15 through end of treatment (24 weeks), 801 mg three times daily
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: Pirfenidone Capsule — Dosing:
  Days 1 through 7, 267 mg three times daily; Days 8 through 14, 534 mg three times daily; Days 15 through end of treatment (24 weeks), 801 mg three times daily duration: 24 weeks
  Other Names: Esbriet
  Arms: Pirfenidone Capsule
Drug: Placebo Capsule — Dosing:
  * Days 1 through 7, 267 mg three times daily;
  * Days 8 through 14, 534 mg three times daily;
  * Days 15 through end of treatment (24 weeks), 801 mg three times daily duration: 24 weeks
  Other Names: Placebo
  Arms: Placebo Capsule

SUMMARY:
Greater than 50% of lung transplant recipients show signs of chronic lung allograft dysfunction (CLAD) by 5 years post-transplantation.Therapies to prevent or slow CLAD are lacking. Anti-fibrotic therapies may offer an avenue to prevent progression of CLAD and prolong allograft survival. This study investigates if Pirfenidone therapy will stabilize lung function decline and slow progression of Functional small airways disease (fSAD) in lung transplant recipients with CLAD.

DETAILED DESCRIPTION:
The study aimed to enroll lung transplant recipients with an established diagnosis of CLAD. The patients were randomized to receive an anti-fibrotic drug Pirfenidone or Placebo pills for 6 month period. High-resolution CT scan of the chest was utilized to measure the primary endpoint of change in functional small airway disease (fSAD). Pulmonary function testing and spirometry were utilized to measure the secondary endpoint of change in FEV1 and FVC.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipients 18 years of age or older
* Greater than 6 months after single or bilateral lung transplantation
* Baseline FEV1 and FVC values (mean of two highest value measured 3 weeks apart) > 50% predicted (to assure viable graft)
* Diagnosis of CLAD (two consecutive spirometric values of FEV1 alone or both FEV1 and FVC < 80% of baseline)

Exclusion Criteria

* Acute Rejection (AR) diagnosis by biopsy in the 28 days prior to enrollment
* Treatment with pulse steroids, Anti-thymocyte Globulin (ATG), extracorporeal photopheresis (ECP), plasmapheresis, or Immunoglobulin therapy aimed at CLAD within the 28 days prior to enrollment
* If the subject is receiving chronic Azithromycin therapy, the dose must be stable for the 28 days prior to enrollment
* Presence of active pulmonary infection at the time of enrollment as determined by an investigator in consultation with the treating pulmonologist
* Diagnosis of bronchial stenosis either a) requiring stenting, or b) thought to be responsible for the spirometric decline by principal investigator
* Abnormal liver function tests (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN), Alkaline phosphatase > 2.5 x ULN, total bilirubin > ULN) or known cirrhosis (>2 times upper limit of normal of AST/ALT/AP)
* Total white blood cell (WBC) < 3.0 K/uL
* Moderate to Severe Renal insufficiency (CrCl <15 mL/min calculated by the Cockcroft-Gault equation)
* Use of any medication known to cause significant interactions with pirfenidone (strong CYP1A2 inhibitors such as Fluvoxamine or Enoxacin or inducers)
* Pregnancy or lactation. Women of child-bearing potential will have a pregnancy test at enrollment and must agree to maintain highly effective contraception with two methods of birth control from the date of consent through the end of the study.
* Tobacco use within 6 months
* History of alcohol abuse in the past 1 year as determined by the treating pulmonologist
* Any condition other than CLAD that will likely result in death in the next 1 year
* Any condition in the judgement of the principal investigator that would preclude participation in this study
* EKG with QTc interval > 500 msec at screening
* Listed for repeat lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vibha Lama, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirfenidone Capsule: Method of Administration: Oral (capsule)
  Dosing:
  * Days 1 through 7, 267 mg three times daily;
  * Days 8 through 14, 534 mg three times daily;
  * Days 15 through end of treatment (24 weeks), 801 mg three times daily
  Pirfenidone Capsule: Dosing:
  Days 1 through 7, 267 mg three times daily; Days 8 through 14, 534 mg three times daily; Days 15 through end of treatment (24 weeks), 801 mg three times daily duration: 24 weeks
- Placebo Capsule: Method of Administration: Oral (capsule)
  Dosing:
  * Days 1 through 7, 267 mg three times daily;
  * Days 8 through 14, 534 mg three times daily;
  * Days 15 through end of treatment (24 weeks), 801 mg three times daily
  Placebo Capsule: Dosing:
  * Days 1 through 7, 267 mg three times daily;
  * Days 8 through 14, 534 mg three times daily;
  * Days 15 through end of treatment (24 weeks), 801 mg three times daily duration: 24 weeks
Period: Overall Study
Arm/Group | Pirfenidone Capsule | Placebo Capsule
Started | 13 | 11
Completed | 8 | 9
Not Completed | 5 | 2
Not completed — Follow up not possible due to COVID restrictions | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirfenidone Capsule | Placebo Capsule | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (11.6) | 57.5 (13.5) | 58.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 3 | 9 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 24
Lung Function FEV 1, FVC, [Mean (Standard Deviation); unit: liters]
  FEV1 | 1.400769 (0.5887057) | 1.410909 (0.4713906) | 1.41 (0.527)
  FVC | 2.544615 (0.8378904) | 2.517273 (0.7226353) | 2.53 (0.77)
CLAD Phenotype [Count of Participants; unit: Participants] — CLAD is Chronic Lung Allograft Dysfunction
  Participants
    FEV1 First Decline | 5 | 4 | 9
    Concurrent FEV1 and FVC Decline | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Functional Small Airways Disease (fSAD) as Measured by Parametric Response Mapping
Description: Evaluate if pirfenidone compared to placebo will stabilize progression of fSAD by comparison of inspiratory and expiratory high resolution computed tomography (HRCT) images through co-registration to provide quantitative measures of fSAD.
Time Frame: Baseline, 24 weeks
Population: Baseline measures taken from all participants. Post treatment percentage measurements taken only from participants who completed the study.
Measure: Mean (Standard Deviation); unit: percentage of change of fsad
Arm/Group | Pirfenidone Capsule | Placebo Capsule
Number analyzed (Participants) | 13 | 11
percentage of change of fsad
  Baseline percentage fSAD | 14.21 (8.80) | 11.90 (13.08)
  Post treatment percentage fSAD: number analyzed (Participants) | 8 | 9
  Post treatment percentage fSAD | 17.10 (6.43) | 10.62 (9.25)
  Net change: number analyzed (Participants) | 8 | 9
  Net change | -5.8620625 (6.636287) | 0.4497328 (10.91197)
Statistical Analysis 1: Comparison: Pirfenidone Capsule vs Placebo Capsule; P-Value provided is for net change only; Test type: Superiority; p = 0.17697507, t-test, 2 sided

2. Secondary Outcome: Change in Forced Expiratory Volume 1 Over 24 Weeks (FEV1)
Description: Measured by spirometry
Time Frame: Baseline, 24 weeks
Population: Baseline measures taken from all participants. Post treatment percentage measurements taken only from participants with available FEV1 results at 24-week mark.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Pirfenidone Capsule | Placebo Capsule
Number analyzed (Participants) | 13 | 11
liters
  Baseline FEV1 | 1.40 (0.59) | 1.41 (0.47)
  24 week FEV1: number analyzed (Participants) | 10 | 10
  24 week FEV1 | 1.36 (0.57) | 1.35 (0.54)
  Change in FEV1: number analyzed (Participants) | 10 | 10
  Change in FEV1 | -0.12 (0.13) | -0.09 (0.30)
Statistical Analysis 1: Comparison: Pirfenidone Capsule vs Placebo Capsule; P-Value provided is for net change only; Test type: Superiority; p = 0.77367872, Welch Two Sample t-test

3. Secondary Outcome: Change in Forced Vital Capacity (FVC) Over 24 Weeks
Description: Measured by spirometry
Time Frame: Baseline, 24 weeks
Population: Baseline measures taken from all participants. Post treatment percentage measurements taken only from participants with available FVC results at 24-week mark.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Pirfenidone Capsule | Placebo Capsule
Number analyzed (Participants) | 13 | 11
liters
  Baseline FVC | 2.54 (0.84) | 2.52 (0.72)
  24-week FVC: number analyzed (Participants) | 10 | 10
  24-week FVC | 2.52 (0.87) | 2.36 (0.86)
  Change in FVC | -0.06 (0.25) | -0.12 (0.40)
Statistical Analysis 1: Comparison: Pirfenidone Capsule vs Placebo Capsule; P-Value provided is for net change only; Test type: Superiority; p = 0.68595748, t-test, 2 sided

4. Secondary Outcome: Number of Adverse Events Related to Study Treatment
Description: Safety of pirfenidone will be measured by adverse events determined to be related to the study drug through review of medical history, physical exam and laboratory findings.
Time Frame: 28 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Pirfenidone Capsule | Placebo Capsule
Number analyzed (Participants) | 13 | 11
Adverse Events
  AE Definitely Related | 0 | 0
  AE Probably Related | 4 | 0
  AE Possibly Related | 15 | 10
  AE Unlikely to be Related | 8 | 10
  AE Definitely Not Related | 1 | 12
Statistical Analysis 1: Comparison: Pirfenidone Capsule vs Placebo Capsule; Test type: Superiority; p = 0.00127634, Fisher Exact

5. Secondary Outcome: Number of Subjects With Treatment Intolerance
Description: Subjects permanently discontinuing study medication before 24 weeks
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone Capsule | Placebo Capsule
Number analyzed (Participants) | 13 | 11
Participants
  Drug Discontinued | 1 | 1
  Drug Not Discontinued, but Held or Dose Reduced | 5 | 3
  Drug Tolerated | 4 | 6
Statistical Analysis 1: Comparison: Pirfenidone Capsule vs Placebo Capsule; Test type: Superiority; p = 0.80904544, Fisher Exact

ADVERSE EVENTS:
Time Frame: 28 weeks from start of treatment
Arm/Group | Pirfenidone Capsule | Placebo Capsule
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 4/11
Other Adverse Events (participants affected / at risk) | 11/13 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone Capsule (N=13) | Placebo Capsule (N=11)
C. difficile colitis (Infections and infestations) | 0 | 1
Respiratory infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone Capsule (N=13) | Placebo Capsule (N=11)
Edema (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Fever (General disorders) | 0 | 1
Headache (General disorders) | 2 | 0
Leukocytosis (General disorders) | 0 | 1
Lightheadedness/syncope (General disorders) | 1 | 0
Myalgias (General disorders) | 1 | 1
Sleep disturbance (General disorders) | 1 | 0
Weight gain (General disorders) | 0 | 1
Belching (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Gastrointestinal upset (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 8 | 2
Liver function test abnormalities (Hepatobiliary disorders) | 0 | 1
Respiratory infection (Infections and infestations) | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Dry eyes (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Facial hair growth (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Salty lips (Skin and subcutaneous tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Overactive bladder (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03473340/Prot_SAP_000.pdf